CLINICAL TRIAL: NCT05057533
Title: Association Between Primary Headaches and Irritable Bowel Syndrome.
Brief Title: Primary Headaches and Irritable Bowel Syndrome.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamal Helmy, Resident doctor, Assiut University
Other Study IDs: Primary Headaches and IBS
Record Dates: First submitted 2021-09-16; First posted 2021-09-27 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Primary Headache Disorder
MeSH Terms: conditions — Headache Disorders, Primary

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: a questionnaire based on Rome IV Diagnostic criteria of IBS — The Rome IV criteria for the diagnosis of IBS require that patients have had recurrent abdominal pain on average at least 1 day per week during the previous 3 months that is associated with two or more of the following
  1. Related to defecation (may be increased or unchanged by defecation)
  2. Associated with a change in stool frequency
  3. Associated with a change in stool form or appearance The Rome IV criteria (May 2016) only require abdominal pain in defining this condition; "discomfort" is no longer a requirement owing to its nonspecificity, and the recurrent abdominal pain. [2] Supporting symptoms include the following:Altered stool frequency Altered stool form Altered stool passage (straining and/or urgency) Mucorrhea Abdominal bloating or subjective distention.

SUMMARY:
To assess the relationship between primary headaches and irritable bowel syndrome

DETAILED DESCRIPTION:
The association between primary headaches and functional gastrointestinal disorders has been confirmed by many clinical observations. In most patients during the attacks of headache, apart from various neurological and vascular symptoms, gastrointestinal disturbances occur . Functional gastrointestinal disorders, such as irritable bowel syndrome (IBS), are reported in primary headache patients in periods between the attacks as well. On the other hand 23-53% of IBS patients have frequent headaches.

Migraine typically presents relapsing episodes of symptoms including headache, nausea, vomiting, sensory hypersensitivity and mood changes that last for hours to days . Similar to migraine, IBS is characterized by recurrent abdominal pain or discomfort with altered gastrointestinal motility and visceral hypersensitivity that returns to normal between attacks . Both pain disorders lack detectable organic causes .

An emerging model of the brain-gut axis was proposed to explain migraine and IBS as a result of a genetically sensitive nervous system that develops hyperexcitability over time as a response to multiple environmental and immunological factors.

Cluster headache (CH) characterized by its distinctive circadian and circannual periodicity, implicating the role of the hypothalamus in its underlying pathophysiology. CH and IBS are featuring recurrent attacks of pain that possess relationships with circadian rhythms and potentially hypothalamic derangements.

Tension headache that's associated with pain in head described as feeling like a tight band around head, also show many similarities with IBS such causes for both are unknown, and some studies suggest a possible link that could shed light on shared genetics of both condition .

ELIGIBILITY:
Inclusion Criteria:

* age more than 18.
* both sex.
* history suggestive of any type of primary headaches.
* accept to participate in the study.

Exclusion Criteria:

* Intake of medications that can aggravate Headache or IBS.
* Presence of neurological disease other than primary headaches.
* Presence of gastrointestinal disease other than IBS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A group of patients attending headache outpatient clinic of Assuit University hospital diagnosed with primary headaches (migraine , tension Headache or cluster headache)according to a questionnaire based on diagnostic criteria established by the International Headache Society will interviewed with a questionnaire based on Rome IV Diagnostic criteria of IBS to detect the prevalence of IBS among patients with primary headaches
Sampling Method: Non-Probability Sample
Enrollment: 197 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-02-01 (Estimated)

PRIMARY OUTCOMES:
Association between primary headaches and irritable bowel syndrome | Basline
  To Detect the prevalence of IBS among patients with primary headaches

SECONDARY OUTCOMES:
Subtypes of primary headachecs and IBS | Basline
  Detect the intimate correlation between each type of primary headaches and IBS

CONTACTS AND LOCATIONS:
Overall Officials: Reda Badry, MD prof, Study Director; Wael Abbas, Study Director
Locations (1):
- Assiut University hospital, Asyut, Egypt

REFERENCES:
- [Background] Soares RL, Moreira-Filho PF, Maneschy CP, Breijao JF, Schmidte NM. The prevalence and clinical characteristics of primary headache in irritable bowel syndrome: a subgroup of the functional somatic syndromes. Arq Gastroenterol. 2013 Oct-Dec;50(4):281-4. doi: 10.1590/S0004-28032013000400008. PMID 24474230
- [Background] Martami F, Ghorbani Z, Abolhasani M, Togha M, Meysamie A, Sharifi A, Razeghi Jahromi S. Comorbidity of gastrointestinal disorders, migraine, and tension-type headache: a cross-sectional study in Iran. Neurol Sci. 2018 Jan;39(1):63-70. doi: 10.1007/s10072-017-3141-0. Epub 2017 Oct 11. PMID 29022143
- [Background] Doulberis M, Saleh C, Beyenburg S. Is there an Association between Migraine and Gastrointestinal Disorders? J Clin Neurol. 2017 Jul;13(3):215-226. doi: 10.3988/jcn.2017.13.3.215. PMID 28748672